CLINICAL TRIAL: NCT00005121
Title: Framingham Heart Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 900
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Cerebrovascular Accident; Hypertension; Heart Failure, Congestive; Peripheral Vascular Diseases; Arterial Occlusive Diseases; Atherosclerosis; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Stroke; Hypertension; Heart Failure; Peripheral Vascular Diseases; Arterial Occlusive Diseases; Atherosclerosis

SUMMARY:
The Framingham Heart Study was initiated to study the factors associated with the development of cardiovascular disease by employing long-term surveillance of an adult population in Framingham, Massachusetts. The Framingham Offspring Study was initiated to assess familial and genetic factors as determinants of coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

The Framingham Heart Study, initiated in 1948, was designed as a longitudinal investigation of constitutional and environmental factors influencing the development of cardiovascular disease in men and women free of these conditions at the outset. The first person was examined in September 1948 and four years later 5,209 persons had received their first examination. The group has now been followed in the Study for twenty-four subsequent biennial examinations. The need for more information arises from the fact that the epidemiology of cardiovascular disease is incompletely known, estimation of risk is imprecise, and the pattern of cardiovascular disease incidence is changing; these changes need to be documented. Changing patterns of cigarette smoking, nutritional habits and exercise patterns as well as changes in other aspects of lifestyle and advances in medical care may all influence future morbidity and mortality rates for cardiovascular disease. New cases of clinically recognizable cardiovascular disease are less predictable in disease free subjects over age 60, and an already large and growing proportion of the total cardiovascular disease events is now first expressed at these ages. Recently available, technologically advanced measurement tools such as echocardiography need to be evaluated as risk assessors in various age groups. Similarly, the predictive efficacy of recently available lipoprotein cholesterol and apoprotein measurements need to be demonstrated for early onset (age less than 60) as well as later onset cardiovascular disease. Thus, as changes in early detection and treatment of cardiovascular disease advance, prospective epidemiology is needed to document the value and impact of these changes in an organized fashion. Finally, the availability of prospective data on two generations adds to the uniqueness of the Framingham Study among ongoing studies of CVD epidemiology. A determination of the extent and mechanisms by which cardiovascular diseases cluster in families is another important goal of the Framingham Study.

In 1982, the National Institute on Aging initiated a study on senile dementia using the Framingham Heart Study cohort. The study was designed to determine morbidity and mortality outcomes among the 160 subjects identified as suffering from dementia at the 15th biennial examination and to determine incidence of senile dementia among those subjects free of dementia at the 15th biennial examination. Outcome of nursing home admissions was also determined in all study participants.

Biennial comprehensive examinations of the Framingham Heart Study cohort have taken place since 1949. Until examination 12, the study was carried out entirely by the NHLBI. After that time, the Boston University Medical Center, in collaboration with, and using facilities and equipment made available by NHLBI, was responsible for the examinations.

DESIGN NARRATIVE:

Biennial examinations are conducted in the surviving original cohort to obtain information on physical activity, blood pressure, diet, body weight, occupational history, psychosocial factors, and personal habits such as smoking. Special tests include electrocardiographic evaluation, exercise stress test, HLA typing, lipoprotein and apoprotein testing, non-invasive assessment of atherosclerosis, fasting blood glucose, lung function testing, B-scan/Doppler of the carotid and or femoral arteries, and clotting or hemostatic measures. Endpoints include coronary heart disease, stroke, hypertension, congestive heart failure, and peripheral arterial disease.

Members of the Offspring Study were examined for the first time between 1971 and 1975, for the second time between 1979 and 1983, for the third time between 1983 and 1987. Examinations consist of a complete physical examination including resting electrocardiogram, medical history, non-invasive cardiovascular examination, lung function assessment, lipoprotein cholesterol and apoprotein measurements, SMA 25, personal history interview, blood cell ion flux measurement, and platelet function and blood clotting factors measurement.

The 27th exam of approximately 400 survivors of the original cohort is complete. The 28th exam has begun and is ahead of schedule. The 7th exam of the Offspring Cohort began in September 1998 and was completed in December 2001 with 3,500 participants examined. The genome scan is complete with approximately 1,800 samples from 336 families. A Genetics Advisory Panel meets regularly to advise NHLBI on the direction of genetic research within the Framingham Study. Analysis of the genetic and nongenetic data is ongoing and extensive covering such areas as the genetics of lipids, lifetime risk of coronary heart disease, trends in events following Q-wave myocardial infarction, factors affecting left ventricular hypertrophy, and the prevalence and determinants of heart valve disorders.

Initiation of the Third Generation Study was announced in November 2001. Beginning in 2002, the Third Generation Study enrolled 3,900 grandchildren of the Framingham Heart Study's original enrollees. Key goals are to identify new risk factors for heart, lung, and blood diseases, identify genes that contribute to good health and to the development of heart, lung, and blood disease, and to develop new imaging tests that can detect very early stages of coronary atherosclerosis in otherwise healthy adults.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1948-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wolf — Boston University

REFERENCES:
- [Derived] Marquardt JP, Tonnesen PE, Mercaldo ND, Graur A, Allaire B, Bouxsein ML, Samelson EJ, Kiel DP, Fintelmann FJ. Subcutaneous and Visceral Adipose Tissue Reference Values From the Framingham Heart Study Thoracic and Abdominal CT. Invest Radiol. 2025 Feb 1;60(2):95-104. doi: 10.1097/RLI.0000000000001104. Epub 2024 Jul 25. PMID 39047288
- [Derived] Wu Y, Chen C, Wei FF, Liang W, Dong Y, Liu C, Choy M, Dong B. Associations between long-term averages of metabolic parameters in adulthood and cardiac structure and function in later life. Hypertens Res. 2024 Feb;47(2):496-506. doi: 10.1038/s41440-023-01475-9. Epub 2023 Oct 19. PMID 37857766
- [Derived] Tonnesen PE, Mercaldo ND, Tahir I, Dietrich AW, Amayri W, Graur A, Allaire B, Bouxsein ML, Samelson EJ, Kiel DP, Fintelmann FJ. Muscle Reference Values From Thoracic and Abdominal CT for Sarcopenia Assessment: The Framingham Heart Study. Invest Radiol. 2024 Mar 1;59(3):259-270. doi: 10.1097/RLI.0000000000001012. Epub 2023 Sep 18. PMID 37725490
- [Derived] Choy M, Huang Y, Peng Y, Liang W, He X, Chen C, Li J, Zhu W, Wei FF, Dong Y, Liu C, Wu Y. Association between epicardial adipose tissue and incident heart failure mediating by alteration of natriuretic peptide and myocardial strain. BMC Med. 2023 Mar 29;21(1):117. doi: 10.1186/s12916-023-02836-4. PMID 36978080
- [Derived] Lai CQ, Parnell LD, Lee YC, Zeng H, Smith CE, McKeown NM, Arnett DK, Ordovas JM. The impact of alcoholic drinks and dietary factors on epigenetic markers associated with triglyceride levels. Front Genet. 2023 Feb 15;14:1117778. doi: 10.3389/fgene.2023.1117778. eCollection 2023. PMID 36873949
- [Derived] Takvorian KS, Wang D, Courchesne P, Vasan RS, Benjamin EJ, Cheng S, Larson MG, Levy D, Ho JE. The Association of Protein Biomarkers With Incident Heart Failure With Preserved and Reduced Ejection Fraction. Circ Heart Fail. 2023 Jan;16(1):e009446. doi: 10.1161/CIRCHEARTFAILURE.121.009446. Epub 2022 Dec 8. PMID 36475777
- [Derived] Lee YC, Christensen JJ, Parnell LD, Smith CE, Shao J, McKeown NM, Ordovas JM, Lai CQ. Using Machine Learning to Predict Obesity Based on Genome-Wide and Epigenome-Wide Gene-Gene and Gene-Diet Interactions. Front Genet. 2022 Jan 3;12:783845. doi: 10.3389/fgene.2021.783845. eCollection 2021. PMID 35047011
- [Derived] Wang K, Liu H. Association between widespread pain and dementia, Alzheimer's disease and stroke: a cohort study from the Framingham Heart Study. Reg Anesth Pain Med. 2021 Oct;46(10):879-885. doi: 10.1136/rapm-2021-102733. Epub 2021 Aug 16. PMID 34400574
- [Derived] Haslam DE, Peloso GM, Guirette M, Imamura F, Bartz TM, Pitsillides AN, Wang CA, Li-Gao R, Westra JM, Pitkanen N, Young KL, Graff M, Wood AC, Braun KVE, Luan J, Kahonen M, Kiefte-de Jong JC, Ghanbari M, Tintle N, Lemaitre RN, Mook-Kanamori DO, North K, Helminen M, Mossavar-Rahmani Y, Snetselaar L, Martin LW, Viikari JS, Oddy WH, Pennell CE, Rosendall FR, Ikram MA, Uitterlinden AG, Psaty BM, Mozaffarian D, Rotter JI, Taylor KD, Lehtimaki T, Raitakari OT, Livingston KA, Voortman T, Forouhi NG, Wareham NJ, de Mutsert R, Rich SS, Manson JE, Mora S, Ridker PM, Merino J, Meigs JB, Dashti HS, Chasman DI, Lichtenstein AH, Smith CE, Dupuis J, Herman MA, McKeown NM. Sugar-Sweetened Beverage Consumption May Modify Associations Between Genetic Variants in the CHREBP (Carbohydrate Responsive Element Binding Protein) Locus and HDL-C (High-Density Lipoprotein Cholesterol) and Triglyceride Concentrations. Circ Genom Precis Med. 2021 Aug;14(4):e003288. doi: 10.1161/CIRCGEN.120.003288. Epub 2021 Jul 16. PMID 34270325
- [Derived] Block RC, Shearer GC, Holub A, Tu XM, Mousa S, Brenna JT, Harris WS, Tintle N. Aspirin and omega-3 fatty acid status interact in the prevention of cardiovascular diseases in Framingham Heart Study. Prostaglandins Leukot Essent Fatty Acids. 2021 Jun;169:102283. doi: 10.1016/j.plefa.2021.102283. Epub 2021 Apr 24. PMID 33964664
- [Derived] Taron J, Lyass A, Mahoney TF, Ehrbar RQ, Vasan RS, D'Agostino RB Sr, Hoffmann U, Massaro JM, Lu MT. Coronary Artery Calcium Score-Directed Primary Prevention With Statins on the Basis of the 2018 American College of Cardiology/American Heart Association/Multisociety Cholesterol Guidelines. J Am Heart Assoc. 2021 Jan 5;10(1):e018342. doi: 10.1161/JAHA.120.018342. Epub 2020 Dec 22. No abstract available. PMID 33348999
- [Derived] Lai CQ, Parnell LD, Smith CE, Guo T, Sayols-Baixeras S, Aslibekyan S, Tiwari HK, Irvin MR, Bender C, Fei D, Hidalgo B, Hopkins PN, Absher DM, Province MA, Elosua R, Arnett DK, Ordovas JM. Carbohydrate and fat intake associated with risk of metabolic diseases through epigenetics of CPT1A. Am J Clin Nutr. 2020 Nov 11;112(5):1200-1211. doi: 10.1093/ajcn/nqaa233. PMID 32930325
- [Derived] McKeown NM, Dashti HS, Ma J, Haslam DE, Kiefte-de Jong JC, Smith CE, Tanaka T, Graff M, Lemaitre RN, Rybin D, Sonestedt E, Frazier-Wood AC, Mook-Kanamori DO, Li Y, Wang CA, Leermakers ETM, Mikkila V, Young KL, Mukamal KJ, Cupples LA, Schulz CA, Chen TA, Li-Gao R, Huang T, Oddy WH, Raitakari O, Rice K, Meigs JB, Ericson U, Steffen LM, Rosendaal FR, Hofman A, Kahonen M, Psaty BM, Brunkwall L, Uitterlinden AG, Viikari J, Siscovick DS, Seppala I, North KE, Mozaffarian D, Dupuis J, Orho-Melander M, Rich SS, de Mutsert R, Qi L, Pennell CE, Franco OH, Lehtimaki T, Herman MA. Sugar-sweetened beverage intake associations with fasting glucose and insulin concentrations are not modified by selected genetic variants in a ChREBP-FGF21 pathway: a meta-analysis. Diabetologia. 2018 Feb;61(2):317-330. doi: 10.1007/s00125-017-4475-0. Epub 2017 Nov 2. PMID 29098321
- [Derived] Fretts AM, Follis JL, Nettleton JA, Lemaitre RN, Ngwa JS, Wojczynski MK, Kalafati IP, Varga TV, Frazier-Wood AC, Houston DK, Lahti J, Ericson U, van den Hooven EH, Mikkila V, Kiefte-de Jong JC, Mozaffarian D, Rice K, Renstrom F, North KE, McKeown NM, Feitosa MF, Kanoni S, Smith CE, Garcia ME, Tiainen AM, Sonestedt E, Manichaikul A, van Rooij FJ, Dimitriou M, Raitakari O, Pankow JS, Djousse L, Province MA, Hu FB, Lai CQ, Keller MF, Perala MM, Rotter JI, Hofman A, Graff M, Kahonen M, Mukamal K, Johansson I, Ordovas JM, Liu Y, Mannisto S, Uitterlinden AG, Deloukas P, Seppala I, Psaty BM, Cupples LA, Borecki IB, Franks PW, Arnett DK, Nalls MA, Eriksson JG, Orho-Melander M, Franco OH, Lehtimaki T, Dedoussis GV, Meigs JB, Siscovick DS. Consumption of meat is associated with higher fasting glucose and insulin concentrations regardless of glucose and insulin genetic risk scores: a meta-analysis of 50,345 Caucasians. Am J Clin Nutr. 2015 Nov;102(5):1266-78. doi: 10.3945/ajcn.114.101238. Epub 2015 Sep 9. PMID 26354543
- [Derived] Cassidy A, Rogers G, Peterson JJ, Dwyer JT, Lin H, Jacques PF. Higher dietary anthocyanin and flavonol intakes are associated with anti-inflammatory effects in a population of US adults. Am J Clin Nutr. 2015 Jul;102(1):172-81. doi: 10.3945/ajcn.115.108555. Epub 2015 May 27. PMID 26016863
- [Derived] Dashti HS, Follis JL, Smith CE, Tanaka T, Cade BE, Gottlieb DJ, Hruby A, Jacques PF, Lamon-Fava S, Richardson K, Saxena R, Scheer FA, Kovanen L, Bartz TM, Perala MM, Jonsson A, Frazier-Wood AC, Kalafati IP, Mikkila V, Partonen T, Lemaitre RN, Lahti J, Hernandez DG, Toft U, Johnson WC, Kanoni S, Raitakari OT, Perola M, Psaty BM, Ferrucci L, Grarup N, Highland HM, Rallidis L, Kahonen M, Havulinna AS, Siscovick DS, Raikkonen K, Jorgensen T, Rotter JI, Deloukas P, Viikari JS, Mozaffarian D, Linneberg A, Seppala I, Hansen T, Salomaa V, Gharib SA, Eriksson JG, Bandinelli S, Pedersen O, Rich SS, Dedoussis G, Lehtimaki T, Ordovas JM. Habitual sleep duration is associated with BMI and macronutrient intake and may be modified by CLOCK genetic variants. Am J Clin Nutr. 2015 Jan;101(1):135-43. doi: 10.3945/ajcn.114.095026. Epub 2014 Nov 26. PMID 25527757
- [Derived] Dashti HS, Shea MK, Smith CE, Tanaka T, Hruby A, Richardson K, Wang TJ, Nalls MA, Guo X, Liu Y, Yao J, Li D, Johnson WC, Benjamin EJ, Kritchevsky SB, Siscovick DS, Ordovas JM, Booth SL. Meta-analysis of genome-wide association studies for circulating phylloquinone concentrations. Am J Clin Nutr. 2014 Dec;100(6):1462-9. doi: 10.3945/ajcn.114.093146. Epub 2014 Oct 8. PMID 25411281
- [Derived] Hunninghake GM, Hatabu H, Okajima Y, Gao W, Dupuis J, Latourelle JC, Nishino M, Araki T, Zazueta OE, Kurugol S, Ross JC, San Jose Estepar R, Murphy E, Steele MP, Loyd JE, Schwarz MI, Fingerlin TE, Rosas IO, Washko GR, O'Connor GT, Schwartz DA. MUC5B promoter polymorphism and interstitial lung abnormalities. N Engl J Med. 2013 Jun 6;368(23):2192-200. doi: 10.1056/NEJMoa1216076. Epub 2013 May 21. PMID 23692170
- [Derived] Tanaka T, Ngwa JS, van Rooij FJ, Zillikens MC, Wojczynski MK, Frazier-Wood AC, Houston DK, Kanoni S, Lemaitre RN, Luan J, Mikkila V, Renstrom F, Sonestedt E, Zhao JH, Chu AY, Qi L, Chasman DI, de Oliveira Otto MC, Dhurandhar EJ, Feitosa MF, Johansson I, Khaw KT, Lohman KK, Manichaikul A, McKeown NM, Mozaffarian D, Singleton A, Stirrups K, Viikari J, Ye Z, Bandinelli S, Barroso I, Deloukas P, Forouhi NG, Hofman A, Liu Y, Lyytikainen LP, North KE, Dimitriou M, Hallmans G, Kahonen M, Langenberg C, Ordovas JM, Uitterlinden AG, Hu FB, Kalafati IP, Raitakari O, Franco OH, Johnson A, Emilsson V, Schrack JA, Semba RD, Siscovick DS, Arnett DK, Borecki IB, Franks PW, Kritchevsky SB, Lehtimaki T, Loos RJ, Orho-Melander M, Rotter JI, Wareham NJ, Witteman JC, Ferrucci L, Dedoussis G, Cupples LA, Nettleton JA. Genome-wide meta-analysis of observational studies shows common genetic variants associated with macronutrient intake. Am J Clin Nutr. 2013 Jun;97(6):1395-402. doi: 10.3945/ajcn.112.052183. Epub 2013 May 1. PMID 23636237
- Available data/document: Individual Participant Data Set: FHS-Cohort — http://biolincc.nhlbi.nih.gov/studies/framcohort/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval, and completion of a data use agreement.
- Available data/document: Study Protocol: FHS-Cohort — http://biolincc.nhlbi.nih.gov/studies/framcohort/
- Available data/document: Study Forms: FHS-Cohort — http://biolincc.nhlbi.nih.gov/studies/framcohort/
- Available data/document: Data Coding Manuals: FHS-Cohort — http://biolincc.nhlbi.nih.gov/studies/framcohort/
- Available data/document: Individual Participant Data Set: FHS-OS — http://biolincc.nhlbi.nih.gov/studies/framoffspring/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval, and completion of a data use agreement.
- Available data/document: Study Protocol: FHS-OS — http://biolincc.nhlbi.nih.gov/studies/framoffspring/
- Available data/document: Study Forms: FHS-OS — http://biolincc.nhlbi.nih.gov/studies/framoffspring/
- Available data/document: Data Coding Manuals: FHS-OS — http://biolincc.nhlbi.nih.gov/studies/framoffspring/
- Available data/document: Individual Participant Data Set: FHS-Gen III — http://biolincc.nhlbi.nih.gov/studies/gen3/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval, and completion of a data use agreement.
- Available data/document: Study Protocol: FHS-Gen III — http://biolincc.nhlbi.nih.gov/studies/gen3/
- Available data/document: Study Forms: FHS-Gen III — http://biolincc.nhlbi.nih.gov/studies/gen3/
- Available data/document: Data Coding Manuals: FHS-Gen III — http://biolincc.nhlbi.nih.gov/studies/gen3/